CLINICAL TRIAL: NCT00384748
Title: Home-Based Tele-Health Stroke Care: A Randomized Trial for Veterans
Brief Title: Home-based Telehealth Stroke Care: A Randomized Trial for Veterans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: B4492-R
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Cerebrovascular Accident
Keywords: Cerebrovascular Accident; Rehabilitation; Telemedicine
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tele-visit Group (Experimental): TR intervention targets safe functional mobility within a home environment and consists of: 1) exercise targeting underlying stroke-related impairment and 2) adaptive strategies targeting external factors to help compensate for disability. TR uses a combination of tele-video visits, an in-home messaging device, and telephone contact over a 3-month study period. A video camera is used in the home to provide visual and audio to a therapist located at the base hospital. An interactive, in-home messaging device is used to facilitate adherence with treatment recommendations and to screen for depression, falls, and difficulty with self-care. This allows evaluations of problem areas during tele-visits, rapid response to new functional problems.
  Interventions: Behavioral: TR intervention; Behavioral: In-home messaging device.
- Usual Care Group (Active Comparator): Patients randomized to the Usual Care group receive routine VA care, as directed by their physicians. Therapy services are tracked via a weekly diary for the entire 6 month study period. In this weekly diary, patients in both the usual care and intervention group will record receipt of therapy. Usual Care group will be asked whether they exercised, and if so how frequently. They will be administered telephone interviews at baseline, 3-and 6-months. The interview outcome measures are FONEFIM, Late-Life Function and Disability Instrument, Falls Self Efficacy Scale and Stroke Specific Patient Satisfaction with Care. In addition, sociodemographics, stroke severity, length of time since stroke onset, and depression at baseline will be measured.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: TR intervention — The 3 tele-visits will occur within 5 weeks post randomization. Telephone call visits will occur during weeks 2, 4, 6, 8 and 12. One additional tele-visit may be scheduled as needed. The first visit is devoted to mobility assessment, goal-setting. The second visit is to review the current exercise component. Visit 3 focuses on functional mobility using adaptive strategy component.
  Other Names: Tele-visit intervention
  Arms: Tele-visit Group
Behavioral: In-home messaging device. — The purpose of this aspect of the intervention is to screen for unforeseen problems and to reinforce adherence to the recommended treatment. It will be used to interface with patients daily, but briefly. The in-home messaging device, which resembles a caller ID box is attached to the home telephone line and electrical outlet. Installation of the equipment involves connecting it to the phone line and plugging it into an electrical outlet. The teletherapist receives the clinical data from the in-home messaging device via the internet on a daily basis. It is used to screen for depression, lower extremity strength, self-care tasks and mobility, falls and exercise adherence.
  Arms: Tele-visit Group
Behavioral: Usual care — Routine VA care.
  Arms: Usual Care Group

SUMMARY:
The purpose of the proposed study is to examine a Tele-rehabilitation (TR) intervention that uses tele-health technology to improve outcomes of stroke patients after discharge to home. The primary aim is to determine the effect of TR on physical function, and secondarily to determine the effect on disability, falls-related self-efficacy, and patient satisfaction.

DETAILED DESCRIPTION:
Stroke patients clearly benefit from intensive, coordinated, inpatient care. At the same time, there is considerable interest in ways to reduce hospital lengths of stay. Early discharge rehabilitation programs require coordinated, well-organized home-based rehabilitation, and lack of sufficient information about the home setting impedes successful rehabilitation. Unfortunately, resources for in-home rehabilitation are limited. The goal of TR is to improve functional mobility using a multifaceted rehabilitation intervention via two types of telehealth technology. Tele-video is used to carry out an in-home assessment of functional mobility, to make treatment recommendations, and to provide periodic goal-oriented reassessment, modifying the treatment plan as the patient improves. Tele-video uses a video camera with a home health aide in the patient's home to provide visual and audio to a therapist located at the base hospital. It is used to carry out an in-home assessment of functional mobility, to make treatment recommendations, and to provide periodic goal-oriented reassessment, modifying the treatment plan as the patient improves. An interactive, in-home messaging device is used to facilitate adherence with treatment recommendations and to screen for interval problems (depression, falls, and difficulty with self-care).

This is a Phase II, 2-arm, 3-site Randomized Controlled Trial (RCT). A total of 120 veterans with recent onset of ischemic or hemorrhagic stroke who are discharged to the community will be randomly assigned to one of two groups: (a) TR; and (b) Usual Care. Dependent variables (physical function, disability, falls-related self-efficacy, and patient satisfaction) will be measured at baseline, 3-, and 6-months via telephone interviews by the study coordinator located at the CIEBP who will be blinded to the study group assignment of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Have acute ischemic or hemorrhagic stroke within the preceding twenty-four months, defined as "a rapid onset event of vascular origin reflecting a focal disturbance of cerebral function, excluding isolated impairments of higher function and persisting longer than 24 hours";
* age between 45-90;
* discharge to the community;
* cognitively intact (score of 6/10 or greater on the Short Portable Mental Status Questionnaire);
* discharge motor Functional Independence Measure (FIM) score of 17-88 (i.e., maximal assistance on no more than 4 motor activities of daily living (ADLs) as the most severe stroke included and modified independence at least 2 motor ADLs as the least severe); able to follow 3-step command; signed VHA Medical Media release form; concurrence by the patient's physician;
* and informed consent

Exclusion Criteria:

Unable to provide informed consent

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neale R. Chumbler, PhD MA BS, Principal Investigator — Richard Roudebush VA Medical Center, Indianapolis; Patricia A Quigley, PhD MPH, Principal Investigator — James A. Haley Veterans Hospital
Locations (3):
- United States (3):
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Medical Center, Durham, Durham, North Carolina

REFERENCES:
- [Result] Lutz BJ, Chumbler NR, Lyles T, Hoffman N, Kobb R. Testing a home-telehealth programme for US veterans recovering from stroke and their family caregivers. Disabil Rehabil. 2009;31(5):402-9. doi: 10.1080/09638280802069558. PMID 18720112
- [Result] Chumbler NR, Rose DK, Griffiths P, Quigley P, McGee-Hernandez N, Carlson KA, Vandenberg P, Morey MC, Sanford J, Hoenig H. Study protocol: home-based telehealth stroke care: a randomized trial for veterans. Trials. 2010 Jun 30;11:74. doi: 10.1186/1745-6215-11-74. PMID 20591171
- [Result] Chumbler NR, Morey M, Quigley P, Rose D, Sanford J, Hoenig H. Tele-rehabilitation for Stroke Care: A Randomized Trial for Veterans. [Abstract]. Telemedicine journal and e-health : the official journal of the American Telemedicine Association. 2010 May 1; 16 Suppl 1:s30.
- [Result] Chumbler NR, Morey MC, Griffiths P, Quigley P, Haley JA, Rose DK, Sanford J, Hoenig H. The Effects of a Stroke Telerehabilitation In-Home Intervention on Function and Disability: Preliminary Results of a Randomized Clinical Trial. [Abstract]. Stroke; A Journal of Cerebral Circulation. 2011 Mar 1; 42(3):e76.
- [Result] Chumbler NR, Quigley P, Li X, Morey M, Rose D, Sanford J, Griffiths P, Hoenig H. Effects of telerehabilitation on physical function and disability for stroke patients: a randomized, controlled trial. Stroke. 2012 Aug;43(8):2168-74. doi: 10.1161/STROKEAHA.111.646943. Epub 2012 May 24. PMID 22627983

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: TR intervention consists of two parts 1) exercise targeting underlying stroke-related impairment and 2) adaptive strategies to help compensate for disability. An in-home messaging device is used to facilitate adherence with treatment recommendations and to screen for problems. This will allow targeted evaluations of problem areas during tele-visits, rapid response to new functional problems.
  The 3 tele-visits will occur within 5 weeks post randomization. Telephone call visits will occur during even weeks.The first visit is devoted to mobility assessment, goal-setting. The second visit is to review the current exercise component. In-home messaging device. The teletherapist receives the clinical data from the in-home messaging device on a daily basis to screen for depression, lower extremity strength, self-care tasks and mobility, falls and exercise adherence.
- Arm 2: Patients randomized to the Usual Care group receive routine VA care, as directed by their physicians.
  Receipt of therapy services will be tracked via a weekly diary for the entire 6 months of the intervention period. In this weekly diary, patients in both the usual care and intervention group will record receipt of therapy. The patients will be asked to include the time in minutes that they spent in receipt of therapy services. Both groups will also be asked whether or not they exercised, and if so how frequently. TR and Usual Care participants will be administered telephone interviews at baseline, 3-and 6-months. The interview outcome measures are FONEFIM, Late-Life Function and Disability Instrument, Falls Self Efficacy Scale and Stroke Specific Patient Satisfaction with Care. In addition, sociodemographics, stroke severity, length of time since stroke onset, and depression at baseline will be measured.
  Usual care: Routine VA care.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 25 | 23
Completed | 25 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Physical Function as Measured by Telephone Version of FIM
Description: The FONEFIM was developed as a telephonic alternative and yields good concordance to the in-person, performance based FIM.12 The motor subscale of the FONEFIM (Motor FONEFIM) consists of 13 items encompassing four categories: 1) self-care; 2) sphincter control; 3) transfers; and 4) locomotion. Each item is scored on an ordinal scale from 1= total dependence to 7 = total independence. Possible scores range from 13 to 91, with higher scores indicating greater independence. The scoring considers the use of adaptive equipment and/or the extent of personal assistance or supervision required to complete the task.
Time Frame: 6-month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 25 | 23
units on a scale | 83.7 (9.9) | 80.9 (12.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the enrollment of the first subject until all subjects had completed the study.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No